CLINICAL TRIAL: NCT00574717
Title: Enhancement of Emmetropization in Hyperopic Infants
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding support for continued recruitment, enrollment, treatment
Sponsor: Ohio State University (Other)
Collaborators: The Ohio Lions Eye Research Foundation (Unknown)
Responsible Party: Principal Investigator, Donald Mutti, Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004H0157
Record Dates: First submitted 2007-12-11; First posted 2007-12-17 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Hyperopia; Hypermetropia; Farsightedness
Keywords: hyperopia; ocular refraction; infant; vision
MeSH Terms: conditions — Hyperopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Infants will receive spectacle under-correction of their hyperopia.
  Interventions: Procedure: Spectacles

INTERVENTIONS:
Procedure: Spectacles — Infants will receive spectacles with 3.00D of under-correction relative to the spherical equivalent in each eye as measured by the cycloplegic retinoscopy performed at baseline. They will also receive the full amount of measured astigmatism in their glasses. Changes in spectacle lens power will be made as needed at follow-up visits to keep the level of under-correction within 0.50D of the target 3.00D. A program of visual engagement is also provided to encourage the normal development and use of accommodation. Treatment will continue for 15 months (until 18 months of age) or until the infant reaches a spherical equivalent refractive error of +3.00D or less hyperopia.
  Other Names: Under-correction

SUMMARY:
To determine if wearing a moderate spectacle under-correction (3.00D) and performing activities designed to stimulate accurate accommodation during a 15-month period will enhance emmetropization in highly hyperopic (between +5.00D and +7.00D) 3-month old infants.

DETAILED DESCRIPTION:
The purpose of the project is to determine if emmetropization can be enhanced in very farsighted babies. We will give them glasses with a partial correction, an amount that is less than their full degree of farsightedness but enough to put them in the zone of effective emmetropization. This 'boost' is meant to enable very farsighted babies to use their eyes in a normal way and emmetropize as normal infants. This partial correction would be given at 3 months of age for a period of up to 15 months. A program of visual engagement is also provided in order to encourage the normal development and use of accommodation. As changes in farsightedness occur, the power of the glasses will be reduced at follow up appointments to keep the farsightedness within the zone of effective emmetropization. Once an infant reaches a normal amount of farsightedness, the glasses would be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* 3 months of age (between 8 weeks and 20 weeks)at the baseline examination
* Either gender, any ethnicity
* Birthweight greater than 2500g
* Normal pregnancy and delivery (including Cesarean section delivery but excluding serious complications or conditions such as eclampsia or rubella)
* Hyperopia of +5.00D or more but less than +7.00D spherical equivalent refractive error in each eye by cycloplegic retinoscopy using cyclopentolate 1%
* Currently under the care of a pediatrician

Exclusion Criteria:

* Anisometropia greater than 1.00D (difference in spherical equivalent)
* Strabismus
* Previous history of difficulty with pupillary dilation
* History of cardiac, liver, asthma, or other respiratory disease
* History of ocular disease or active ocular inflammation

Ages: 8 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be to determine if the criterion level for emmetropization (≤+3.00D by 18 months of age) is met and maintained by at least 70% of treated infants. | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald O. Mutti, OD, PhD, Principal Investigator — The Ohio State University College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

REFERENCES:
- [Background] Atkinson J, Anker S, Bobier W, Braddick O, Durden K, Nardini M, Watson P. Normal emmetropization in infants with spectacle correction for hyperopia. Invest Ophthalmol Vis Sci. 2000 Nov;41(12):3726-31. PMID 11053269
- [Background] Ingram RM, Gill LE, Lambert TW. Effect of spectacles on changes of spherical hypermetropia in infants who did, and did not, have strabismus. Br J Ophthalmol. 2000 Mar;84(3):324-6. doi: 10.1136/bjo.84.3.324. PMID 10684846
- [Background] Mutti DO, Mitchell GL, Jones LA, Friedman NE, Frane SL, Lin WK, Moeschberger ML, Zadnik K. Axial growth and changes in lenticular and corneal power during emmetropization in infants. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3074-80. doi: 10.1167/iovs.04-1040. PMID 16123404
- [Background] Mutti DO, Mitchell GL, Jones LA, Friedman NE, Frane SL, Lin WK, Moeschberger ML, Zadnik K. Refractive astigmatism and the toricity of ocular components in human infants. Optom Vis Sci. 2004 Oct;81(10):753-61. doi: 10.1097/00006324-200410000-00007. PMID 15557849
- [Background] Anker S, Atkinson J, Braddick O, Nardini M, Ehrlich D. Non-cycloplegic refractive screening can identify infants whose visual outcome at 4 years is improved by spectacle correction. Strabismus. 2004 Dec;12(4):227-45. doi: 10.1080/09273970490517935. PMID 15545141
- [Background] Hung LF, Crawford ML, Smith EL. Spectacle lenses alter eye growth and the refractive status of young monkeys. Nat Med. 1995 Aug;1(8):761-5. doi: 10.1038/nm0895-761. PMID 7585177
- [Background] Schaeffel F, Glasser A, Howland HC. Accommodation, refractive error and eye growth in chickens. Vision Res. 1988;28(5):639-57. doi: 10.1016/0042-6989(88)90113-7. PMID 3195068
- [Background] Smith EL 3rd, Hung LF. The role of optical defocus in regulating refractive development in infant monkeys. Vision Res. 1999 Apr;39(8):1415-35. doi: 10.1016/s0042-6989(98)00229-6. PMID 10343811
- See also: College of Optometry Website — http://optometry.osu.edu/?n=0
- See also: Principal Investigator Web Page — http://optometry.osu.edu/directory/faculty_detail.cfm?id=mutti.2